# Clinical Development and Regulatory Affairs Biostatistics and Data Management



## STATISTICAL ANALYSIS PLAN

| Title: | A PHASE 3, DOUBLE-MASKED, RANDOMIZED STUDY OF THE EFFICACY AND SAFETY OF INTRAVITREAL AFLIBERCEPT INJECTION IN PATIENTS WITH MODERATELY SEVERE TO SEVERE NONPROLIFERATIVE DIABETIC RETINOPATHY |
|---|---|
| Protocol: | VGFTe-OD-1411 |
| Investigational product: | Intravitreal Aflibercept Injection |
| Sponsor: | Regeneron Pharmaceuticals, Inc. |
| Study Biostatistician: | |
| Clinical Trial Manager: | |
| Study Medical Director: | |
| Date: | 09 July 2018 |

3.0

Version:

The approval signatures below indicate that these individuals have reviewed the Statistical Analysis Plan (SAP) and agreed on the planned analysis defined in this document for reporting.

See appended electronic signature page

I Approve this Document

Study Biostatistician

See appended electronic signature page

I Approve this Document

Study Medical Director

See appended electronic signature page

I Approve this Document

Head of BDM or designee

## TABLE OF CONTENTS

| LIST OF | F ABBREVIATIONS AND DEFINITION OF TERMS | 6 |
|---|---|---|
| DOCUM | MENT VERSION HISTORY | 8 |
| 1. | OVERVIEW | 9 |
| 1.1. | Background/Rationale | 9 |
| 1.2. | Study Objectives | 10 |
| 1.2.1. | Primary Objectives | 10 |
| 1.2.2. | Secondary Objectives | 10 |
| 1.2.3. | Modifications from the Statistical Section in the Final Protocol | 10 |
| 1.2.4. | Modifications from the Approved Statistical Analysis Plan | 10 |
| 2. | INVESTIGATION PLAN | 11 |
| 2.1. | Study Design and Randomization | 11 |
| 2.2. | Sample Size and Power Considerations | 12 |
| 3. | ANALYSIS POPULATIONS | 13 |
| 3.1. | Full Analysis Set | 13 |
| 3.2. | Safety Analysis Set | 13 |
| 3.3. | Subgroup Analysis Set | 13 |
| 4. | ANALYSIS VARIABLES | 15 |
| 4.1. | Demographic and Baseline Characteristics | 15 |
| 4.2. | Medical History | 15 |
| 4.3. | Pre-Treatment / Concomitant Medication | 15 |
| 4.4. | Exposure, Compliance, Additional Treatment to Study Treatment | 16 |
| 4.5. | Efficacy Variable | 16 |
| 4.5.1. | Primary Efficacy Variable (s) | 16 |
| 4.5.2. | Secondary Efficacy Variable(s) | 16 |
| 4.5.3. | Additional Efficacy Variable(s) | 17 |
| 4.6. | Safety Variables | 18 |
| 4.6.1. | Adverse Events and Serious Adverse Events | 18 |
| 4.6.2. | Surgeries | 19 |
| 4.6.3. | Laboratory Safety Variables | 19 |
| 4.6.4. | Vital Signs | 19 |
| 4.6.5. | 12-Lead Electrocardiography (ECG) | 19 |

| 4.6.6. | Ocular Safety Measures | 20 |
|---|---|---|
| 5. | STATISTICAL METHODS | 21 |
| 5.1. | Statistical Hypothesis | 21 |
| 5.2. | Demographics, Baseline Characteristics, Medical History, and Prior/<br>Concomitant Medication | 22 |
| 5.3. | Subject Disposition | 22 |
| 5.4. | Extent of Study Treatment Exposure and Compliance | 23 |
| 5.5. | Analyses of Efficacy Variables | 23 |
| 5.5.1. | Analysis of Primary Efficacy Variable(s) | 23 |
| 5.5.1.1. | Primary Analysis for Primary Efficacy Variable | 23 |
| 5.5.1.2. | Sensitivity Analyses for Primary Efficacy Variable | 24 |
| 5.5.2. | Analysis of Secondary Efficacy Variables | 25 |
| 5.5.3. | Analysis of Additional Efficacy Variables | 26 |
| 5.5.4. | Subgroup Analyses | 26 |
| 5.6. | Analysis of Safety Data | 26 |
| 5.6.1. | Adverse Events | 27 |
| 5.6.2. | Surgeries | 27 |
| 5.6.3. | Clinical Laboratory | 27 |
| 5.6.4. | Vital Signs | 28 |
| 5.6.5. | Electrocardiogram | 28 |
| 5.6.6. | Ocular Safety Measures | 28 |
| 6. | DATA CONVENTIONS | 29 |
| 6.1. | Definition of Baseline | 29 |
| 6.2. | Unscheduled Assessments | 29 |
| 6.3. | Subset of Week 24 and Week 52 Analysis Windows | 29 |
| 6.4. | Handling of Patients who Discontinue | 29 |
| 6.5. | Handling of Missing Data | 30 |
| 6.5.1. | General Rules | 30 |
| 7. | INTERIM ANALYSIS | 31 |
| 8. | SOFTWARE | 31 |
| 9. | REFERENCES | 31 |
| 10. | APPENDIX | 32 |
| 10.1. | Schedule of Time and Events: | 32 |

| 10.2. | Summary of Statistical Efficacy Analyses | 37 |
|---|---|---|
| 10.3. | Detailed Definition of Selected Subgroups | 39 |
| 10.3.1. | Hypertension | 40 |
| 10.3.2. | Medical history of Cerebrovascular accident (CVA) / Stroke | 41 |
| 10.3.3. | Medical history of ischemic heart disease /Myocardial Infarction: defined by MSSO SMO 20000047 | 46 |
| 10.3.4. | Renal Impairment | 51 |
| 10.4. | Calculation of confidence intervals using Mantel-Haenszel weighting scheme | 52 |
| 10.5. | Criteria for Predefined Lab Abnormalities | 53 |
| 10.6. | Process to Derive Week 24 (Week 52) Data Cut-off | 55 |
| 10.6.1. | Visit Dependent Data | 55 |
| 10.6.2. | Visit Independent Data | 55 |
| 10.6.3. | Study Medication Data | 56 |
| 10.7. | SAS Procedure for Multiple Imputation | 57 |
| | LIST OF TABLES | |
| Table 1: | Significance Levels for Testing Secondary Efficacy Endpoints | 21 |
| | LIST OF FIGURES | |
| Figure 1: | Study Flow Diagram | 12 |

#### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AE Adverse Event

ALT Alanine Aminotransferase

ASNV Anterior segment neovascularization

AST Aspartate Aminotransferase

ATC Anatomical Therapeutically Chemical

AUC Area Under the Curve

BCVA Best Corrected Visual Acuity

BUN Blood Urea Nitrogen
CI-DME Central-Involved DME
CMH Cochran-Mantel-Haenszel

CRF Case Report Form

DME Diabetic Macular Edema

DRSS Diabetic Retinopathy Severity Score

ETDRS Early Treatment Diabetic Retinopathy Study

FA Fluorescein Angiography

FAS Full Analysis Set

FP Fundus Photography

IAI Intravitreal Aflibercept Injection

ICF Informed Consent Form

ICH International Conference of Harmonization

IOP Intraocular Pressure

IVRS Interactive Voice Response System

IWRS Interactive Web Response System

IVT Intravitreal

LDH Lactate Dehydrogenase

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

(MedDRA) HLT High Level Term (MedDRA) LLT Low Level Term (MedDRA) PT Preferred Term

(MedDRA) SOC System Organ Class

NPDR Nonproliferative Diabetic Retinopathy

OCT Optical Coherence Tomography

PPS Per Protocol Set

PDR Proliferative Diabetic Retinopathy

PRP Panretinal Photocoagulation

RBC Red Blood Cell

SAE Serious Adverse Event

SAF Safety Analysis set

SAP Statistical Analysis Plan

SD-OCT Spectral Domain Optical Coherence Tomography

TEAE Treatment-emergent Adverse Event

UPCR Urine protein creatinine ratio

VA Visual Acuity

VEGF Vascular Endothelial Growth Factor

WBC White Blood Cell

WHO World Health Organization

## **DOCUMENT VERSION HISTORY**

| Version | Date | Version History |
|---|---|---|
| 1.0 | 21DEC2015 | Initial Version |
| 2.0 | 17FEB2016 | Purpose: Update to incorporate the following revisions in response to feedback from the Food and Drug Administration (FDA) and the Pharmaceuticals and Medical Devices Agency (PMDA): |
| | | 1. Revise the significance levels for testing of the secondary efficacy endpoints in Table 1 of Section 5.1, per FDA feedback |
| | | Add multiple imputation SAS code in Appendix 10.7 per FDA feedback |
| | | 3. Add a hemoglobin A1c assessment at week 24, and fundus photography at week 8 in Appendix 10.1, per PMDA feedback |
| 3.0 | 09JUL2018 | Purpose: Change the timepoint for evaluation of the secondary endpoints from week 100 to week 52. Changes may be found in Section 1, Figure 1 of Section 2.1, Section 4.5.2, Section 4.5.3, Section 5.1, Section 5.5, Section 5.5.2, Section 5.5.3 and Appendix 10.2 |

#### 1. **OVERVIEW**

The purpose of the statistical analysis plan (SAP) is to ensure the credibility of the study results by pre-specifying the statistical approaches for the analysis of the study. The statistical evaluation will be done according to the specifications given in the protocol and, if applicable, the corresponding amendments.

The SAP is intended to be a comprehensive and detailed description of the strategy and statistical technique to be used for the analysis of Week 24 (Visit 7), Week 52 (Visit 11), and Week 100 (Visit 18) data from the VGFTe-OD-1411 study. The statistical analysis of the Week 24 and Week 52 (the primary timepoints) data will be performed as soon as the Week 24 and Week 52 data of all patients are available, even though the study will be ongoing.

This SAP covers the following three analyses:

- Analysis of the data through Week 24 as primary analysis for combined 2Q8 and 2Q16 groups (only data from the combined treatment group and the sham group will be summarized)
- Analysis of the data up to Week 52 as primary and secondary analysis for 2Q8 and 2Q16 groups separately
- Analysis of all endpoints in an exploratory manner at Week 100 for all 3 groups

## 1.1. Background/Rationale

Diabetes mellitus and its complications are a worldwide health epidemic that is expected to increase. In 2013, the World Health Organization (WHO) estimated that 347 million people had diabetes and this number has been projected to increase to 366 million by 2030 and potentially more if rates of obesity continue to increase. Despite early intervention programs and better methods of glycemic control, morbidity and mortality as a consequence of diabetes, including diabetic retinopathy, are expected to rise. Diabetic retinopathy is microvascular damage to the blood vessels in the retina, and it can progress to vision-threatening stages including proliferative diabetic retinopathy (PDR), where new vessels that are susceptible to hemorrhage grow initially from the retina and/or optic disc and extend beyond the internal limiting membrane, and diabetic macular edema (DME), where fluid accumulates disrupting the macular architecture and function. Although there are treatments for DME (eg, anti-vascular endothelial growth factor [VEGF] agents), there is a significant unmet medical need for the treatment of diabetic retinopathy. More advanced retinopathy (proliferative) is often treated with panretinal photocoagulation (PRP). Although PRP may stop the progression of a proliferative disease, it is inherently destructive to the retina and, therefore, likely to cause visual symptoms such as visual field defects, reduced contrast sensitivity, and impaired night and color vision, and can also lead to exacerbation of macular edema. There is currently no treatment for nonproliferative diabetic retinopathy (NPDR), and patients are observed until disease progresses sufficiently to warrant PRP.

Intravitreal (IVT) anti-VEGF therapy is currently the standard of care treatment for DME, and it has proven to be generally safe and effective in patients with DME. In the phase 3 VISTA and VIVID studies of EYLEA® (aflibercept, known in the scientific literature and in clinical studies as VEGF Trap-Eye or intravitreal aflibercept injection [IAI]), patients treated with either

aflibercept 2 mg every 4 weeks (2Q4) or aflibercept 2 mg every 8 weeks (2Q8) (following 5 initial monthly doses) regimens gained 11.5 and 10.7 letters, respectively, in best corrected visual acuity (BCVA) at week 52.

Despite advances in treatment for DME, there are currently no approved treatments for NPDR in patients without DME, leaving patients at risk for the development of PDR and/or DME. Based on the evidence from the VISTA and VIVID studies in patients with DME showing that EYLEA (in addition to treating macular edema) also improves the underlying diabetic retinopathy, we propose to investigate EYLEA in patients with moderately severe to severe NPDR who do not have DME by assessing the proportion of patients who improve by at least 2 steps on the DRSS (Diabetic Retinopathy Severity Score).

This phase 3 study will assess the efficacy and safety of IVT aflibercept in patients with moderately severe to severe NPDR.

## 1.2. Study Objectives

## 1.2.1. Primary Objectives

The primary objective of the study is to assess the efficacy of IVT aflibercept compared to sham treatment in the improvement of moderately severe to severe NPDR.

## 1.2.2. Secondary Objectives

The secondary objectives of the study are:

- To characterize the safety of IVT aflibercept in patients with moderately severe to severe NPDR
- To determine if IVT aflibercept will prevent the worsening of diabetic retinopathy and reduce the incidence of DME
- To determine the anatomic effects of IVT aflibercept in patients with moderately severe to severe NPDR

#### 1.2.3. Modifications from the Statistical Section in the Final Protocol

Not applicable

#### 1.2.4. Modifications from the Approved Statistical Analysis Plan

Not applicable

#### 2. INVESTIGATION PLAN

## 2.1. Study Design and Randomization

This is a phase 3, double-masked, randomized study of the efficacy and safety of IVT aflibercept for the improvement of moderately severe to severe NPDR.

After providing informed consent, patients will be assessed for study eligibility at the screening visit, up to 3 weeks before day 1/baseline. At the day 1/baseline visit, patients will undergo safety assessments prior to receiving the first dose of study drug.

Eligible patients will be enrolled into 1 of 3 treatment groups in a 1:1:1 randomization scheme, and will be stratified based on their DRSS score (level 47 vs. level 53). Only 1 eye will be selected as the study eye. The 3 treatment groups will have the following dosing regimens from day 1 to week 48: 1) 2Q8 aflibercept IVT after 5 initial monthly doses; 2) 2Q16 aflibercept IVT after 3 initial monthly doses and one 8-week interval; and 3) sham treatment. In year 2 (beginning at week 56), the 2Q8 group will be treated with a flexible treatment regimen.

The primary outcome measure of the study is the proportion of patients who have improved by ≥2 steps from baseline on the DRSS in the combined 2Q8 and 2Q16 groups at week 24, and in each group individually at week 52. Patients will be evaluated for efficacy (BCVA using the 4-meter ETDRS (Early Treatment Diabetic Retinopathy Study) protocol, spectral domain optical coherence tomography [SD-OCT], and fluorescein angiography [FA]/fundus photography [FP]) and for ocular and systemic safety (including ophthalmic exams, visual field testing, and laboratory assessments) through week 100 (Figure 1).

Patients who develop PDR, anterior segment neovascularization (ASNV), or DME will qualify for rescue treatment. If treatment is given, subsequent patient data will be censored for the primary analysis.

Figure 1: Study Flow Diagram



Approximately 360 patients will be randomized in a 1:1:1 ratio to receive either aflibercept 2Q8, aflibercept 2Q16, or sham according to a central randomization scheme provided by an interactive voice response system (IVRS)/interactive web response system (IWRS) to the designated study pharmacist (or qualified designee). Randomization will be stratified according to the patient's DRSS level (level 47 vs. level 53 at the screening visit).

The study event table is presented in Appendix 10.1.

## 2.2. Sample Size and Power Considerations

Anticipating approximately 41% of patients with a  $\geq$ 2-step improvement from baseline in DRSS score at week 52 in either the 2Q8 or 2Q16 groups versus 17% in the sham group, 102 patients per group are required to detect a difference with a power of 90% for rejecting the null hypothesis at a 2-sided 1.67% (5%/3) significance level. A sample size of 102 patients per group will provide at least 90% power to detect a difference between combined aflibercept group vs. sham group at week 24, if a 38% response rate is assumed in the combined aflibercept group. The assumption of the proportions for the aflibercept group and sham group is based on VIVID and VISTA data at a given time point. To account for about a 15% dropout rate, 120 patients per group will be enrolled.

The sample size calculation was computed using the Chi square test (continuity corrected) from the commercial software nQuery nTerm 7.0.

#### 3. ANALYSIS POPULATIONS

In accordance with guidance from the International Conference of Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) guideline ICH E9 Statistical Principles for Clinical Trials (1998), the following analysis populations will be used for all statistical analysis:

## 3.1. Full Analysis Set

<u>The full analysis set (FAS)</u> includes all randomized patients who received any study treatment. Analysis of the FAS will be performed according to the treatment assigned at baseline (as randomized). The efficacy analysis on the FAS is considered to be the primary one (statistical evaluation of superiority). The FAS will be used to evaluate all efficacy endpoints for Week 24, Week 52 and Week 100 data.

## 3.2. Safety Analysis Set

<u>Safety analysis set (SAF)</u> includes all randomized patients who receive at least 1 study treatment (aflibercept or sham). Patients will be summarized according to the treatment actually received (as treated). The 'as-treated' assignment will only differ from the "as randomized" if the patient is systematically receiving treatment from an alternative treatment group. However, isolated incorrect treatments will not constitute a change in the "as treated" assignment. Patients whose "as treated" assignment differs from their "as randomized" assignment will be listed.

Treatment administration/ compliance, all clinical safety, and tolerability assessments will be analyzed using the SAF for Week 24, Week 52 and Week 100 data. The safety analysis will be performed on the observed safety data.

## 3.3. Subgroup Analysis Set

Subgroups are defined by key baseline factors recorded on the case report form (CRF) and listed as follows:

- Subgroups to be considered for both efficacy and safety analyses
  - 1. Sex
  - 2. Age: <40y; >=40-<65y; >=65y
  - 3. Race: White, Black or African American, Other
  - 4. Ethnicity: Hispanic or Latino (no/yes)
  - 5. HbA1C:  $\leq 8\%$ ; > 8%

- Subgroups to be considered for efficacy analyses only
  - 1. Baseline DRSS score: 47 vs. 53
- Subgroups to be considered for safety analyses only
  - 1. Medical history of hypertension
  - 2. Medical history of cerebrovascular disease (e.g., CVA/stroke)
  - 3. Medical history of ischemic heart disease (e.g., myocardial infarction)
  - 4. Renal impairment

- Normal: > 80 ml/min

- Mild: > 50-80 ml/min

- Moderate: > 30-50 ml/min

- Severe: <= 30 ml/min or requiring dialysis

CrCl is calculated according Cockcroft-Gault formula (renal impairment guideline of FDA, 1998):

$$CrCl \approx \frac{[140 - age(years)] * weight(kg)}{72 * serum creatinine(mg/dl)} * \begin{cases} 1.0, if male \\ 0.85, if female \end{cases}$$

Subjects are considered requiring dialysis if their medical history includes one of preferred terms (PTs).

The detailed definition of the PTs for the safety subgroups above is presented in Appendix 10.3.

#### 4. ANALYSIS VARIABLES

## 4.1. Demographic and Baseline Characteristics

Demographic and baseline assessments to be summarized will include:

- Age, gender, and race
- Age category: <40y; >=40-<65y; >=65y
- Weight, height, BMI (kg/m²)
- Smoking history
- HbA1C
- HbA1C category: <= 8%; >8%
- BMI  $\leq 30 \text{ kg/m}^2$ , BMI  $\geq 30 \leq 35 \text{ kg/m}^2$ , BMI  $\geq 35 \text{ kg/m}^2$
- Vital Signs (Baseline heart rate, systolic blood pressure, diastolic blood pressure and temperature)
- Baseline Intraocular pressure (IOP)
- Medical History
- Duration of Diabetes (years): defined as time from diagnosis (based on medical history data (MedDRA HLT "diabetes mellitus") to randomization
- Diabetes Type (Type 1 and Type 2)
- Baseline DRSS
- Baseline ETDRS letter score
- Baseline central retinal thickness

## 4.2. Medical History

Medical history will be coded according to latest available version of Medical Dictionary for Regulatory Activities (MedDRA).

## 4.3. Pre-Treatment / Concomitant Medication

Medications taken during the study will be recorded and will be coded to ATC codes according to the World Health Organization Drug Dictionary (WHO Drug Dictionary) 2005Q3 enhanced version provided by Bayer Health Care.

Mediations will be summarized as follows:

- **Prior medication** is defined as medication that was started before and ended before a patient received first study treatment (active or sham treatment)
- **Concomitant medication** is defined as medications that are ongoing at, or begin after the start of study treatment

• **New medication** is defined as medications that began after the start of study treatment

The prior, concomitant and new medication will be summarized by ATC class (ATC level 1) and subclass (ATC level 2).

Variables for concomitant medication description and analysis will include Generic name, ATC level codes, Indication, Dose/Dose Unit, Frequency, Route, start/end date and study day, Duration, Ongoing.

## 4.4. Exposure, Compliance, Additional Treatment to Study Treatment

## **Exposure**

For each patient, the following variables will be used to examine exposure to study treatment for the study eye (rescue treatment will not be taken into account here:

- Total number of active injections in aflibercept groups
- Total number of sham injections separately by treatment groups
- Duration of treatment calculated (Weeks) as: [(last study treatment date) (first study treatment date) + 28]/7 (28 days are added because of the minimum 4-week dosing interval in the study)
- For patients who receive rescue treatment for PDR, ASNV, or CI-DME, the type, frequency and duration of treatment will be summarized

#### **Compliance**

Per patient, compliance with protocol-defined study medication during the time periods: 24 weeks, 52 weeks and 100 weeks will be calculated as follows:

Treatment Compliance =

(Number of received injections [sham or active] through week time period)/(Number of planned injections [sham or active] during period of participation in the study through time period) x 100%

For the calculation of compliance all injections (regardless if they were sham or active) will be used

## 4.5. Efficacy Variable

## 4.5.1. Primary Efficacy Variable (s)

The primary efficacy variable is the proportion of patients who have improved by  $\ge 2$  steps from baseline in the DRSS score at week 24 in the combined 2Q8 and 2Q16 groups and at week 52 for the separate groups.

#### 4.5.2. Secondary Efficacy Variable(s)

The secondary outcome measures will be tested at week 52 and are as follows:

• Proportion of patients developing a vision-threatening complication due to diabetic retinopathy

Vision-threatening complications are defined as composite outcome of PDR (inclusive of patients who have vitreous hemorrhage or tractional retinal detachment believed to be due to PDR) and ASNV

Note: ASNV is defined as neovascularization of the iris (at least 2 cumulative clock hours), and/or definitive neovascularization of the iridocorneal angle

- Proportion of patients who develop central-involved DME (CI-DME)
- Time to development of a vision-threatening complication
- Time to development of CI-DME
- Proportion of patients who receive PRP, inclusive of patients undergoing vitrectomy with endolaser
- Area under the curve (AUC) for change in BCVA from baseline

## 4.5.3. Additional Efficacy Variable(s)

The additional outcome measures in the study are:

- Time to first improvement of ≥2 steps from baseline in the DRSS score through week 52 and week 100
- Proportion of patients with ≥2-step improvement from baseline in the DRSS score at week 100
- Proportion of patients with ≥2-step worsening from baseline in the DRSS score at week 52 and at week 100
- Proportion of patients with ≥3-step worsening from baseline in the DRSS score at week 52 and at week 100
- Proportion of patients with ≥3-step improvement from baseline in the DRSS score at week 52 and at week 100
- Proportion of patients who receive vitrectomy through week 52 and through week 100
- Change in central retinal thickness from baseline at week 52 and at week 100
- Change in mean deviation on visual field testing from baseline at week 52 and at week 100
- Change in BCVA from baseline at week 24, week 52 and week 100
- Proportion of patients who have gained ≥5, ≥10, or ≥15 letters from baseline at week 52 and at week 100
- Proportion of patients who have lost  $\geq 5$ ,  $\geq 10$ , or  $\geq 15$  letters from baseline at week 24, week 52 and week 100

- The proportion of patients who are equal to or better than 20/20 or equal to or better than 20/40 at week 52 and at week 100.
- Proportion of patients developing either a vision-threatening complication or CI-DME through week 100
- Time to development of either a vision-threatening complication or CI-DME through week 100

## Secondary Endpoints to be tested as Exploratory

- Proportion of patients developing a vision-threatening complication through week 100
- Proportion of patients who develop CI-DME through week 100
- Time to development of a vision-threatening complication through week 100
- Time to development of CI-DME through week 100
- Proportion of patients who receive PRP through week 100, inclusive of patients undergoing vitrectomy with endolaser
- Area under the curve (AUC) for change in BCVA from baseline through week 24 and 100

## 4.6. Safety Variables

#### 4.6.1. Adverse Events and Serious Adverse Events

An adverse event (AE) is any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug.

Adverse events will be collected at each visit from the time of informed consent signature until the end of the study. If the patient withdraws from the study during the screening, AEs will be collected up until the patient withdraws. If the patient withdraws at any point after receiving the first dose of study medication, AEs will be collected up until 30 days after the last dose of study drug or the termination visit, whichever is later.

Adverse events will be summarized as:

- **Pre-treatment AE:** Include adverse events that occur after the patient has signed the informed consent, but prior to Visit 2 (Day 1, date of the patient's first dose of study drug).
- Treatment-Emergent Adverse Event (TEAE): TEAE is defined as AE that is observed or reported after first and not later than 30 days after last administration of study medication (active or sham injection) or aflibercept injection in the fellow eye. Only worsening, pre-existing AEs and new AEs reported during treatment period (period after first treatment) will be collected in the study.

The following study periods will be used for TEAE and AE summaries:

• Day 1 to Week 24

- Day 1 to Week 52
- Day 1 to Week 100, End of Study

The data cut-off rules for Week 24 and Week 52 AE reporting are described in Appendix 10.6.

Other variables for AE description and analysis will include AE Verbatim Term, AE start date and end date/ongoing and corresponding study day, AE Duration, relationship of AE to study drug, relationship of AE to study procedure, seriousness, intensity, action due to AE, treatment of AE and outcome.

#### 4.6.2. Surgeries

All the surgeries after informed consent are collected on the CRF and are coded by MedDRA. The following variables will be tabulated by MedDRA preferred term:

- Pre-treatment surgery is defined as surgery performed before the start of study treatment (active or sham)
- Treatment emergent surgery is defined as surgery performed on or after the start of study treatment (active or sham)
  - Ocular treatment emergent surgery for study eye and fellow eye
  - Non-ocular treatment emergent surgery

#### 4.6.3. Laboratory Safety Variables

Clinical laboratory variables will include the following:

- Blood chemistry panel: Sodium, Potassium, Chloride, Carbon dioxide, Calcium, Glucose, Albumin, Total Protein, serum, Creatine, Blood urea nitrogen (BUN), Aspartate, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase, Lactate dehydrogenase (LDH), Total bilirubin, Total cholesterol, Uric acid, Creatine phosphokinase
- Hematology panel: Hemoglobin, Hematocrit, Red blood cells (RBC), White blood cells (WBC), Red Cell Indices, Platelet count, Differential count: Neutrophils, Lymphocytes, Monocytes, Basophils, Eosinophils
- Urinalysis: Color, Clarity, pH, Specific gravity, Ketones, Protein, Urine protein creatinine ratio (UPCR), Glucose, Blood, Blood, Bilirubin, Leukocyte esterase, Nitrite, WBC, RBC, Hyaline and other casts, Bacteria, Epithelial cells, Crystals, Yeast, Creatinine
- Hemoglobin A1c, Vitamin D

#### 4.6.4. Vital Signs

Variables of analysis for vital signs include temperature, heart rate and blood pressure measures.

#### 4.6.5. 12-Lead Electrocardiography (ECG)

12-Lead ECG parameters include

ECG variables will include heart rate, PR interval, RR interval, QRS duration, QT interval, overall interpretation of ECG (normal/abnormal) and clinically relevant abnormalities (no/yes). QTc with Bazett and Fridericia correction will be calculated.

## 4.6.6. Ocular Safety Measures

Variables of analysis for ocular safety measures include during Week 24, Week 52 and Week 100:

- Proportion of patient with increased intraocular ocular pressure (IOP)
  - ≥ 10 mmHg increase in IOP measurement from baseline to any pre-dose measurement
  - > 21 mmHg for any pre-dose measurement
  - $\geq$  25 mmHg for any pre-dose measurement
  - $\geq 35$  mmHg at any time

Post dose IOP measurement should be the last IOP recorded.

#### 5. STATISTICAL METHODS

All efficacy and safety variables will be summarized descriptively with appropriate statistics: categorical variables by frequency (absolute and relative frequencies) and continuous variables by sample statistics (i.e. mean, standard deviation, minimum, median, quartiles and maximum). Continuous variables will be described by visit and as change from Baseline, if applicable.

## 5.1. Statistical Hypothesis

This study will examine the following hypotheses for the primary efficacy variable regarding the proportion of patients with a ≥2-step improvement from baseline in DRSS score in the study eye at week 24 in the combined 2Q8 and 2Q16 groups, and at week 52 for the 2Q8 and 2Q16 groups individually. Statistical testing of week 24 and week 52 will be conducted to demonstrate the superiority of the aflibercept groups (combined, 2Q8 and 2Q16) to the sham group, respectively.

For each test, let  $p_t$  (and  $p_c$ ) be the true proportion of patients with a  $\geq$ 2-step improvement from baseline in DRSS score at week 24 for the combined 2Q8 and 2Q16 groups, and at week 52 for the 2Q8 and 2Q16 groups individually (and the sham group,  $p_c$ ).

The following hypotheses will be tested:

$$H_0$$
:  $p_t = p_c$  versus  $H_1$ :  $p_t \neq p_c$ 

To control the family-wise type I error rate of 5%, primary efficacy endpoints for the combined group (week 24) and endpoints for the 2Q8 and 2Q16 groups (week 52) will be tested separately at the significance level of  $\alpha = 1.67\%$  (5%/3). Secondary efficacy endpoints at week 52 will be tested for 2Q8 and 2Q16 groups by the hierarchical testing procedure at a significance level based on values in Table 1 for different scenarios with the predefined testing order.

**Table 1:** Significance Levels for Testing Secondary Efficacy Endpoints

| Scenario | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Combined Group at Week 24 Positive? | X | X | X | | X | | |
| 2Q8 Group at Week 52 Positive? | X | X | | X | | X | |
| 2Q16 Group at Week 52<br>Positive? | X | | X | X | | | X |
| Significance level for secondary endpoints | 0.05 | 0.033 | 0.033 | 0.033 | | 0.0167 | 0.0167 |
| Significance level for Testing for 2Q8 Group at week 52 | 0.025 | 0.033 | | 0.0167 | | 0.0167 | |
| Significance level for Testing for 2Q16 at week 52 | 0.025 | | 0.033 | 0.0167 | | | 0.0167 |

## **5.2.** Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medication

Demographic data and baseline characteristics variables described in Section 4.1 will be summarized using descriptive statistics for SAF and FAS.

Medical history is evaluated for SAF by a frequency table, showing number of patients with medical history findings by primary system organ class (SOC), high level term (HLT) by MedDRA terms.

Prior/concomitant medication will be summarized by WHO-DD 2005Q3 enhanced version ATC codes (ATC 3-digit class and ATC 5-digit subclass) for medication taken during the study. Separate frequency tables will be displayed for patients with prior medications, new medications and concomitant medications by the time periods described in Section 4.3.

Concomitant medications will be summarized by the following periods:

- Day 1 up to Week 24
- Day 1 up to Week 52
- Day 1 up to End of study

## 5.3. Subject Disposition

The following categories for patient disposition will be summarized descriptively:

- The total number of screened patients: met the inclusion criteria regarding the target indication and signed the informed consent form (ICF)
- The total number and percentage of randomized patients: received a randomization number
- The number and percentage of patients in each analysis set
- The total number and percentage of patients who discontinued the study at Week 24, Week 52 and Week 100 with the reasons for discontinuation

The following listings will be provided to assess the patient disposition:

- A listing of patients treated but not randomized and patients randomized but not treated if any
- A listing of patients who developed a vision threatening complication or central-involved DME through week 52 and through week 100
- A listing of patients who received rescue treatment in the study eye
- A listing of patients who were withdrawn from the study, along with reasons for discontinuation
- Listing of major protocol deviations: violation of inclusion/exclusion criteria; post-enrollment deviations which will impact assessment of efficacy endpoints

## 5.4. Extent of Study Treatment Exposure and Compliance

The variables for dose exposure and compliance described in Section 4.4 will be summarized for study eye in SAF and FAS population, using descriptive statistics by the following time periods:

- Day 1 to Week 24 (excluding treatment at Week 24)
- Day 1 to Week 52
- Day 1 to Week 100

## 5.5. Analyses of Efficacy Variables

Efficacy analyses of all efficacy variables defined in Section 4.5 will be conducted using the FAS population.

The primary endpoint analysis for the study will be conducted at 2 time points (week 24 for the combined 2Q8 and 2Q16 groups and week 52 for the 2Q8 and 2Q16 groups individually). Each of the primary efficacy analyses will be tested at the 1.67% (5%/3) significance level to control for multiplicity.

The secondary endpoints described in Section 4.5.2 for 2Q8 and 2Q16 groups will be tested separately in a hierarchical manner at week 52 as described in Section 5.1.

#### 5.5.1. Analysis of Primary Efficacy Variable(s)

## 5.5.1.1. Primary Analysis for Primary Efficacy Variable

The primary analysis is a statistical evaluation of superiority of 3 comparisons (combined aflibercept vs. sham at week 24, aflibercept 2Q8 vs. sham at week 52, and aflibercept 2Q16 vs. sham at week 52) in respect to the primary efficacy variable (see Section 4.5.1). The statistical analysis will be performed using the Cochran-Mantel-Haenszel (CMH) method, stratified by baseline DRSS level (level 47 vs. level 53). Missing or non-gradable post-baseline values will be imputed using the last observation carry forward (LOCF) procedure. For any patient who receives rescue treatment, measurements after rescue is given will be imputed using the last observation prior to rescue treatment. Baseline will be carried forward if all post-baseline observations are missing or non-gradable.

Patients will be considered as non-responders if baseline observations are missing or non-gradable.

Aflibercept treatment will be considered to be superior to sham if the estimated aflibercept group (combined, aflibercept 2Q8, or aflibercept 2Q16) is greater than the sham group, and the p-value is less than or equal to or statistically significant at a 1.67% level.

## 5.5.1.2. Sensitivity Analyses for Primary Efficacy Variable

The following sensitivity analyses are used for the primary efficacy variable:

• Observed case (OC) analysis

Measurements taken after the initiation of rescue treatment will be censored; only observed, gradable, and non-censored values will be used for analysis, (i.e. missing or non-gradable data will not be imputed).

Patients who have received rescue treatment

In these analyses the value at the given timepoint will be used regardless of whether the patient received rescue treatment or not. Two different analyses will be conducted:

- Ancillary LOCF (aLOCF) Data obtained after the initiation of rescue treatment will be included; missing or non-gradable data will be imputed by LOCF.
   Baseline will be carried forward if all post-baseline observations are missing or non-gradable. The data will be analyzed in the same way as described for the primary analysis in Section 5.5.1.1.
- Ancillary observed case (aOC) All observed values will be used for analysis, including measurements taken after the initiation of rescue treatment is given.
   Missing or non-gradable data will not be imputed. The data will be analyzed in the same way as described for the primary analysis in Section 5.5.1.1.
- Multiple imputation

The primary efficacy variable will also be analyzed by multiple imputation on FAS. Multiple imputation method will be conducted by the following three steps:

- a. Imputation Missing or non-gradable DRSS data will be imputed using MI procedure based on the observed case (OC) data. First, missing data will be imputed to achieve a monotone missing pattern using the MCMC (Markov Chain Monte Carlo) method with number of imputations = 100. Subsequently missing data will be imputed by a regression model with number of imputation = 1.
- b. Analysis The responder variable which is the improvement at least 2-step in DRSS can be determined from the complete DRSS data sets. The proportion of the responder will be analyzed using Cochran-Mantel-Haenszel test with stratification adjustment for baseline DRSS level (level 47 vs. level 53).
- c. Pooling Cochran-Mantel-Haenszel statistic from step b, under the null hypothesis, has an asymptotic chi-square distribution. It will be transformed to standard normal distribution by Wilson-Hilferty transformation. After normalization, the analysis results from multiple imputed data sets will be combined into one overall result based on Rubin's rules using MIANALYZE procedure.

SAS procedure for multiple imputation is described in Appendix 10.7.

## 5.5.2. Analysis of Secondary Efficacy Variables

If at least one of the aflibercept groups is shown to be superior to sham in the primary variable, additional comparisons will be made for this aflibercept group with respect to the secondary variables at week 52 with the specified significance level as described in Section 5.1.

A hierarchical testing procedure will be performed for each dose group to compare the secondary variables between the respective aflibercept group and sham in the following order:

- 2Q8 secondary endpoints at week 52
  - Proportion of patients developing a vision-threatening complication
  - Proportion of patients who develop CI-DME
  - Time to development of a vision-threatening complication
  - Time to development of CI-DME
  - Proportion of patients who receive PRP, inclusive of patients undergoing vitrectomy with endolaser
  - Area under the curve (AUC) for change in BCVA from baseline
- 2Q16 secondary endpoints at week 52
  - Proportion of patients developing a vision-threatening complication
  - Proportion of patients who develop CI-DME
  - Time to development of a vision-threatening complication
  - Time to development of CI-DME
  - Proportion of patients who receive PRP, inclusive of patients undergoing vitrectomy with endolaser
  - Area under the curve (AUC) for change in BCVA from baseline

The p-values at week 52 for the secondary endpoints will be reported for all comparisons between the aflibercept groups and the sham group; however, a superiority claim can be made for a given endpoint only if all preceding endpoint comparisons in the hierarchy are shown to be statistically significant at the significance level specified in Section 5.1. The hierarchical method ensures the overall type I error rate of 5% for this study, with multiplicity adjustment for primary and secondary endpoint analyses.

All endpoints will also be analyzed descriptively at week 100 in an exploratory manner.

The analysis of proportion variables will be done using the same methodology as for the analyses of the primary efficacy variable described in Section 5.5.1.

For continuous variables (ie, BCVA), an analysis of covariance (ANCOVA) model with baseline measurements of the continuous variable as covariates and treatment and baseline DRSS score (level 47 vs. level 53) stratification as fixed factors will be used for the endpoint. The pair-wise comparisons of each aflibercept group versus sham will be done in the ANCOVA model. In

addition, 2-sided 95% confidence intervals for the difference of each aflibercept group minus sham will be calculated.

Time to first vision-threatening complication will be analyzed using the Kaplan-Meier estimates. A log-rank test will be performed, comparing sham with the aflibercept groups, as well as 2-sided 95% confidence intervals for the time to first vision-threatening complication for the difference of each comparison group. Time to development of CI-DME will be analyzed similarly.

Similar to the analysis of the primary endpoint, missing or non-gradable post-baseline values will be imputed using the last observation carry forward (LOCF) procedure. Baseline will be carried forward if all post-baseline observations are missing. The following sensitivity analyses will be done for secondary efficacy endpoints: OC, aLOCF, and aOC as defined in Section 5.5.1.2.

### 5.5.3. Analysis of Additional Efficacy Variables

All additional efficacy variables (see Section 4.5.3) will be analyzed descriptively. The p-values in the analysis will be nominal and only for descriptive purpose. In addition, the primary and secondary variables will also be analyzed descriptively as additional variables at week 100. These descriptive analyses may include statistical tests on the proportion for the efficacy variables, in the same way as described for the primary and secondary efficacy variable analyses (see Section 5.5.1 and Section 5.5.2).

The analysis of categorical variables will be done using the same methodology used for the analysis of the primary efficacy variable described in Section 5.5.1. Analyses of continuous variables (eg, central retinal thickness, median deviation on visual field) will use a 2-way ANCOVA main effects models with treatment group and baseline DRSS (level 47 vs. level 53) stratification as fixed factors and respective baseline value for the efficacy measure in question as a covariate. The pairwise comparisons of each aflibercept treatment group versus sham will be done in these models by corresponding CONTRAST statements and a point-estimate. A 2-sided 95% confidence interval for the treatment difference of each aflibercept treatment group minus sham will be calculated. The analysis of time to event variables will be done using the same method as that described for the time to first vision-threatening complication in Section 5.5.2.

#### 5.5.4. Subgroup Analyses

Subgroup analyses will be performed on the FAS population using descriptive statistics for primary and secondary efficacy variables with LOCF, OC, aLOCF, and aOC methods based on the subgroup variables defined in Section 4.5.

## 5.6. Analysis of Safety Data

The safety variables as described in Section 4.6 will be analyzed on SAF population through Week 24, Week 52 and Week 100 after final study database lock.

#### **5.6.1.** Adverse Events

AE summaries will be constructed displaying frequencies and proportions of patients reporting AEs within each SOC in decreasing order of total frequency according to the numbers of patients reporting the SOC and the AE within the SOC (not number of reports).

AEs will be classified as Pre-treatment AEs and TEAEs, and will further be summarized by the following categories:

- Ocular AEs in the study eye
- Ocular AEs in the fellow eye
- Non-ocular AEs

Serious Adverse Events (SAEs), drug-related AEs, drug-related SAEs, and TEAEs leading to discontinuation will be summarized in the same way as described for TEAE.

TEAEs in the study eye related to the injection procedure and those related to the study medication will be summarized separately.

An overall summary of the AE profile for aflibercept in this study will be provided. A listing will be constructed that includes the patient identification, the treatment group, category of AE (ocular study eye or fellow eye, non-ocular), AE, MedDRA term, seriousness, severity, causality, elapsed time to onset, duration, and outcome.

Adjudicated APTC events, intraocular inflammation, and hypertension will be tabulated and listed.

Subgroup analyses in TEAE reporting will be performed for the subgroups described in Section 3.3, for each of the following types of TEAE:

Summaries (by SOC and PT) of patients with:

- Ocular TEAEs study eye
- Non-ocular TEAEs
- Serious ocular TEAEs study eye
- Serious non-ocular TEAEs

#### 5.6.2. Surgeries

An overall summary of number of patients undergoing surgery as described in Section 4.6.2 through the end of Week 24, Week 52 and Week 100 will be given by treatment group.

#### 5.6.3. Clinical Laboratory

Baseline clinical laboratory values and change from Baseline to each scheduled assessment visit in clinical laboratory variables described in Section 4.6.3 will be summarized using descriptive statistics

Predefined lab abnormalities will be identified for selected clinical laboratory values according to the specified ranges (see Appendix 10.5). The frequency and percentage of subjects with at

least one predefined lab abnormalities during treatment period will be displayed by treatment group for each analytic. Shift tables will also be provided.

Lab values out of normal range will be flagged in lab value listings.

#### 5.6.4. Vital Signs

Baseline vital signs and change from Baseline for vital sign variables described in Section 4.6.4 at each scheduled assessment visit will be summarized using descriptive statistics. These will include the number of patients, mean, median, standard deviation, minimum, and maximum.

## 5.6.5. Electrocardiogram

All ECG variables as described in Section 4.6.5 will be analyzed by appropriate descriptive methods and change from baseline or frequency tables and/or cross-tabulation of baseline vs. post-baseline status for categorical variables (overall interpretation of ECG normal/abnormal and clinical relevant abnormalities no/yes) by visit and treatment arms.

#### **5.6.6.** Ocular Safety Measures

Baseline IOP and change from Baseline in IOP to each scheduled assessment visit will be summarized with descriptive statistics for study eye and fellow eye. Assessment of significant values or increases will be made and summarized for the proportion of patients with increased IOP in the study eye or fellow eye with the categories defined in Section 4.6.6.

#### 6. DATA CONVENTIONS

The following analysis conventions will be used in the statistical analysis.

#### **6.1.** Definition of Baseline

Unless otherwise specified, the Baseline assessment for all measurements will be the last available valid measurement taken prior to the administration of investigational product.

#### **6.2.** Unscheduled Assessments

Assessments taken outside of protocol allowable windows will be displayed according to the case report form (CRF) assessment recorded by the investigator.

Unscheduled and extra assessments (e.g., laboratory data or vital signs associated with non-protocol clinic visits or obtained in the course of investigating or managing adverse events) will be included in listings, but not summaries with the exception of the tabulation of incidence rates (e.g. of lab abnormalities or predefined IOP increases) using all documented values post baseline

If more than one value is available for a given visit, the visit value actually used for statistical summaries and analyses will be as follows:

- The last non-missing repeated measurement, if respective visit is before start of treatment
- First non-missing repeated measurement, if respective visit is after start of treatment

Early termination visit (ET): If a subject prematurely discontinues they are asked to come for an early termination visit. Visit based information of this visit will only be used in the tabulation and in the statistical analyses if the visit was performed 4 weeks (+/- 1 week) after the last scheduled visit. ET visits outside this window will not be used for analyses and handled in the same way as unscheduled assessments (see above) and the data will only be shown in the patient listings.

## 6.3. Subset of Week 24 and Week 52 Analysis Windows

All relevant Week 24 and Week 52 data will be kept in a separate database for the Week 24 and Week 52 analyses, respectively. In the Appendix 10.6, a detailed process to derive the Week 24 and Week 52 cut-off data from the global study is provided.

## 6.4. Handling of Patients who Discontinue

Patients who discontinue this study will not be replaced. The details for the handling of missing data due to patients who discontinue the study and study medication are described in Section 6.5.1.

## 6.5. Handling of Missing Data

#### 6.5.1. General Rules

When appropriate, the following rules will be implemented so as not to exclude patients from statistical analyses due to missing or incomplete data:

## • Efficacy Variables

For the primary, secondary and additional efficacy variables, missing observations will be imputed using LOCF. The details are described in the efficacy analysis section (see Section 5.5).

#### AE variables

For some AEs it is important to determine whether the AE started before or after the first active aflibercept injection. If the AE start date is partially missing, it will be imputed by the latest possible date (considering other available data, e.g., stop date) to be conservative.

#### • Prior/concomitant medication

For the tabulation of prior and concomitant medication, partially missing start dates of the medication will be imputed by the earliest possible time point, partially missing stop dates will be imputed by the latest possible time point.

## 7. INTERIM ANALYSIS

No formal interim analysis is planned.

## 8. SOFTWARE

All analyses will be done using SAS Version 9.2 or higher.

## 9. REFERENCES

ICH. (1998, February 5). ICH Harmonized tripartite guideline: Statistical principles for clinical trials (E9). International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use.

## 10. APPENDIX

## 10.1. Schedule of Time and Events:

Schedule of Events (Year 1)

Visual field testing (study eye)<sup>8</sup>
Non-Ocular Assessments
Physical examination
Vital signs <sup>11</sup>
ECG
Adverse events <sup>12</sup>

<sup>11.</sup> Vital signs (body temper:

<sup>12.</sup> Adverse events will be a withdraws from the study

<sup>13.</sup> All samples collected for

At visits at which FA is 1 be tested at visit 1 (screen

<sup>15.</sup> Sampling only for HbA1

Schedule of Events (Year 2)

childbearing potential<sup>13</sup> Anti-aflibercept antibody samples<sup>14</sup>

- 1. Patients who are withdr
- 2. Patients will receive eitl
- 3. Gonioscopy in the study

be tested at visit 18 (weel

- All women of childbeari required before treatment
- 14. All ADA samples must b
10.2. Summary of Statistical Efficacy Analyses

| Endpoint | | Week<br>52 | 1 | Major<br>Analysis, | Statistical Analysis | Subgroup<br>Analysis | Sensitivity<br>Analysis |
|---|---|---|---|---|---|---|---|
| | | | | population | | | |
| Proportion of patients who have improved by ≥2 steps from baseline in the DRSS score at week 24 in the combined group, and at week 52 for the 2Q8 and 2Q16 groups individually | X | X | X* | LOCF, FAS | Superiority of VEGF<br>aflibercept over Sham<br>using CMH test<br>adjusted by stratifying<br>factor DRSS level | LOCF,<br>OC,<br>aLOCF,<br>aOC in<br>FAS | Multiple<br>imputation,<br>OC,<br>aLOCF,<br>aOC |
| Proportion of patients developing a vision-threatening complication through week 52 | | X | X* | LOCF, FAS | Superiority of<br>aflibercept over Sham<br>using CMH test<br>adjusted by stratifying<br>factor DRSS level | LOCF,<br>OC,<br>aLOCF,<br>aOC in<br>FAS | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients who develop CI-DME through week 52 | | X | X* | LOCF, FAS | Superiority of<br>aflibercept over Sham<br>using CMH test<br>adjusted by stratifying<br>factor DRSS level | LOCF,<br>OC,<br>aLOCF,<br>aOC in<br>FAS | OC,<br>aLOCF,<br>aOC, |
| Time to development of a vision-threatening complication through week 52 | | X | X* | LOCF, FAS | Kaplan-Meier method<br>and logrank test of<br>aflibercept over Sham | | OC,<br>aLOCF,<br>aOC, |
| Time to development of CI-DME through week 52 | | X | X* | LOCF, FAS | Kaplan-Meier method<br>and logrank test of<br>aflibercept over Sham | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients who receive PRP through week 52, inclusive of patients undergoing vitrectomy with endolaser | | X | X* | LOCF, FAS | Superiority of<br>aflibercept over Sham<br>using CMH test<br>adjusted by stratifying<br>factor DRSS level | LOCF,<br>OC,<br>aLOCF,<br>aOC in<br>FAS | OC,<br>aLOCF,<br>aOC, |
| AUC for change in BCVA from baseline at week 52 | X* | X | X* | LOCF, FAS | Test for superiority of<br>aflibercept over Laser<br>using ANCOVA | LOCF,<br>OC,<br>aLOCF,<br>aOC in<br>FAS | OC,<br>aLOCF,<br>aOC, |

| Endpoint | Week<br>24 | Week<br>52 | Week<br>100 | Major<br>Analysis,<br>population | Statistical Analysis | Subgroup<br>Analysis | Sensitivity<br>Analysis |
|---|---|---|---|---|---|---|---|
| Time to first improvement of ≥2 steps from baseline in the DRSS score through week 52 and week 100 | | X* | X* | LOCF, FAS | Kaplan-Meier method | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients with ≥2-step improvement from baseline in the DRSS score at week 100 | | | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients with ≥2-step worsening from baseline in the DRSS score at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients with ≥3-step worsening from baseline in the DRSS score at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients with ≥3-step improvement from baseline in the DRSS score at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients who receive vitrectomy through week 52 and through week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Change in central retinal thickness from baseline at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Change in mean deviation<br>on visual field testing from<br>baseline at week 52 and at<br>week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Change in BCVA from baseline at week 24, week 52 and week 100 | X* | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |

| Endpoint | Week<br>24 | Week<br>52 | Week<br>100 | Major<br>Analysis,<br>population | Statistical Analysis | Subgroup<br>Analysis | Sensitivity<br>Analysis |
|---|---|---|---|---|---|---|---|
| Proportion of patients who have gained ≥5, ≥10, or ≥15 letters from baseline at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients who have lost $\geq 5$ , $\geq 10$ , or $\geq 15$ letters from baseline at week 24, week 52 and at week 100 | X* | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| The proportion of patients who are equal to or better than 20/20 or equal to or better than 20/40 at week 52 and at week 100 | | X* | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Proportion of patients<br>developing a<br>vision-threatening<br>complication or CI-DME<br>through week 100 | | | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |
| Time to development of vision-threatening complication or CI-DME through week 100 | | | X* | LOCF, FAS | Descriptive statistics | | OC,<br>aLOCF,<br>aOC, |

<sup>\*</sup>As additional endpoints (exploratory)

## 10.3. Detailed Definition of Selected Subgroups

In the following the definitions for subgroups based on medical history are given. All PTs given are based on MedDRA version 16.0 and might be updated with the latest version used in the studies.

### 10.3.1. Hypertension

HT defined by selected PT of MSSO SMQ 20000147: 'Hypertension' (these selected PT form the PBMQ)

| MSSO SMQ | MSS SMQ CODE | Preferred term |
|--------------|--------------|----------------------------------------|
| Hypertension | 20000147 | Accelerated hypertension |
| Hypertension | 20000147 | Blood pressure ambulatory increased |
| Hypertension | 20000147 | Blood pressure diastolic increased |
| Hypertension | 20000147 | Blood pressure inadequately controlled |
| Hypertension | 20000147 | Blood pressure increased |
| Hypertension | 20000147 | Blood pressure systolic increased |
| Hypertension | 20000147 | Diastolic hypertension |
| Hypertension | 20000147 | Endocrine hypertension |
| Hypertension | 20000147 | Essential hypertension |
| Hypertension | 20000147 | Hypertension |
| Hypertension | 20000147 | Hypertension neonatal |
| Hypertension | 20000147 | Hypertensive angiopathy |
| Hypertension | 20000147 | Hypertensive cardiomegaly |
| Hypertension | 20000147 | Hypertensive cardiomyopathy |
| Hypertension | 20000147 | Hypertensive crisis |
| Hypertension | 20000147 | Hypertensive emergency |
| Hypertension | 20000147 | Hypertensive encephalopathy |
| Hypertension | 20000147 | Hypertensive heart disease |
| Hypertension | 20000147 | Hypertensive nephropathy |
| Hypertension | 20000147 | Labile hypertension |
| Hypertension | 20000147 | Malignant hypertension |
| Hypertension | 20000147 | Malignant hypertensive heart disease |
| Hypertension | 20000147 | Malignant renal hypertension |
| Hypertension | 20000147 | Maternal hypertension affecting foetus |
| Hypertension | 20000147 | Mean arterial pressure increased |
| Hypertension | 20000147 | Neurogenic hypertension |
| Hypertension | 20000147 | Orthostatic hypertension |
| Hypertension | 20000147 | Prehypertension |
| Hypertension | 20000147 | Renal hypertension |
| Hypertension | 20000147 | Renovascular hypertension |
| Hypertension | 20000147 | Retinopathy hypertensive |
| Hypertension | 20000147 | Systolic hypertension |

10.3.2. Medical history of Cerebrovascular accident (CVA) / Stroke

| 10.3.2. Medic | al history of Cerebrovascular accident (CVA) / Stroke |
|---------------|-------------------------------------------------------|
| SMQ Code | Preferred term |
| 20000060 | Agnosia |
| 20000060 | Amaurosis fugax |
| 20000060 | Amyloid related imaging abnormalities |
| 20000060 | Angiogram cerebral abnormal |
| 20000060 | Aphasia |
| 20000060 | Balint's syndrome |
| 20000060 | Basal ganglia haemorrhage |
| 20000060 | Basal ganglia infarction |
| 20000060 | Basal ganglia stroke |
| 20000060 | Basilar artery occlusion |
| 20000060 | Basilar artery stenosis |
| 20000060 | Basilar artery thrombosis |
| 20000060 | Blood brain barrier defect |
| 20000060 | Brachiocephalic artery occlusion |
| 20000060 | Brain hypoxia |
| 20000060 | Brain injury |
| 20000060 | Brain stem haematoma |
| 20000060 | Brain stem haemorrhage |
| 20000060 | Brain stem infarction |
| 20000060 | Brain stem ischaemia |
| 20000060 | Brain stem microhaemorrhage |
| 20000060 | Brain stem stroke |
| 20000060 | Brain stem thrombosis |
| 20000060 | Capsular warning syndrome |
| 20000060 | Carotid aneurysm rupture |
| 20000060 | Carotid angioplasty |
| 20000060 | Carotid arterial embolus |
| 20000060 | Carotid arteriosclerosis |
| 20000060 | Carotid artery aneurysm |
| 20000060 | Carotid artery bypass |
| 20000060 | Carotid artery disease |
| 20000060 | Carotid artery dissection |
| 20000060 | Carotid artery insufficiency |
| 20000060 | Carotid artery occlusion |
| 20000060 | Carotid artery restenosis |

| SMQ Code | Preferred term |
|----------|--------------------------------------------------|
| 20000060 | Carotid artery stenosis |
| 20000060 | Carotid artery stent insertion |
| 20000060 | Carotid artery stent removal |
| 20000060 | Carotid artery thrombosis |
| 20000060 | Carotid endarterectomy |
| 20000060 | Carotid revascularisation |
| 20000060 | Central nervous system haemorrhage |
| 20000060 | Central pain syndrome |
| 20000060 | Cerebellar artery occlusion |
| 20000060 | Cerebellar artery thrombosis |
| 20000060 | Cerebellar embolism |
| 20000060 | Cerebellar haematoma |
| 20000060 | Cerebellar haemorrhage |
| 20000060 | Cerebellar infarction |
| 20000060 | Cerebellar ischaemia |
| 20000060 | Cerebellar microhaemorrhage |
| 20000060 | Cerebral amyloid angiopathy |
| 20000060 | Cerebral aneurysm ruptured syphilitic |
| 20000060 | Cerebral arteriosclerosis |
| 20000060 | Cerebral arteriovenous malformation haemorrhagic |
| 20000060 | Cerebral arteritis |
| 20000060 | Cerebral artery embolism |
| 20000060 | Cerebral artery occlusion |
| 20000060 | Cerebral artery stenosis |
| 20000060 | Cerebral artery thrombosis |
| 20000060 | Cerebral circulatory failure |
| 20000060 | Cerebral gas embolism |
| 20000060 | Cerebral haematoma |
| 20000060 | Cerebral haemorrhage |
| 20000060 | Cerebral haemorrhage foetal |
| 20000060 | Cerebral haemorrhage neonatal |
| 20000060 | Cerebral haemosiderin deposition |
| 20000060 | Cerebral hypoperfusion |
| 20000060 | Cerebral infarction |
| 20000060 | Cerebral infarction foetal |
| 20000060 | Cerebral ischaemia |

| SMQ Code | Preferred term |
|----------|--------------------------------------------|
| 20000060 | Cerebral microangiopathy |
| 20000060 | Cerebral microhaemorrhage |
| 20000060 | Cerebral revascularisation |
| 20000060 | Cerebral septic infarct |
| 20000060 | Cerebral small vessel ischaemic disease |
| 20000060 | Cerebral thrombosis |
| 20000060 | Cerebral vasoconstriction |
| 20000060 | Cerebral venous thrombosis |
| 20000060 | Cerebrovascular accident |
| 20000060 | Cerebrovascular accident prophylaxis |
| 20000060 | Cerebrovascular arteriovenous malformation |
| 20000060 | Cerebrovascular disorder |
| 20000060 | Cerebrovascular insufficiency |
| 20000060 | Cerebrovascular stenosis |
| 20000060 | Charcot-Bouchard microaneurysms |
| 20000060 | Congenital cerebrovascular anomaly |
| 20000060 | Congenital hemiparesis |
| 20000060 | CSF bilirubin positive |
| 20000060 | Diplegia |
| 20000060 | Dural fistula |
| 20000060 | Dysarthria |
| 20000060 | Embolic cerebral infarction |
| 20000060 | Embolic stroke |
| 20000060 | Extradural haematoma |
| 20000060 | Fahr's disease |
| 20000060 | Foetal cerebrovascular disorder |
| 20000060 | Haemorrhage intracranial |
| 20000060 | Haemorrhagic cerebral infarction |
| 20000060 | Haemorrhagic stroke |
| 20000060 | Haemorrhagic transformation stroke |
| 20000060 | Hemiparesis |
| 20000060 | Hemiplegia |
| 20000060 | Hypoxic-ischaemic encephalopathy |
| 20000060 | Inner ear infarction |
| 20000060 | Internal carotid artery kinking |
| 20000060 | Intra-cerebral aneurysm operation |

| SMQ Code | Preferred term |
|----------|-------------------------------------------|
| 20000060 | Intracerebral haematoma evacuation |
| 20000060 | Intracranial aneurysm |
| 20000060 | Intracranial haematoma |
| 20000060 | Intracranial venous sinus thrombosis |
| 20000060 | Intraventricular haemorrhage |
| 20000060 | Intraventricular haemorrhage neonatal |
| 20000060 | Ischaemic cerebral infarction |
| 20000060 | Ischaemic stroke |
| 20000060 | Lacunar infarction |
| 20000060 | Lateral medullary syndrome |
| 20000060 | Meningorrhagia |
| 20000060 | Millard-Gubler syndrome |
| 20000060 | Modified Rankin score decreased |
| 20000060 | Modified Rankin score increased |
| 20000060 | Monoparesis |
| 20000060 | Monoplegia |
| 20000060 | Moyamoya disease |
| 20000060 | NIH stroke scale abnormal |
| 20000060 | NIH stroke scale score decreased |
| 20000060 | NIH stroke scale score increased |
| 20000060 | Paralysis |
| 20000060 | Paralysis flaccid |
| 20000060 | Paraparesis |
| 20000060 | Paraplegia |
| 20000060 | Paresis |
| 20000060 | Post procedural stroke |
| 20000060 | Post stroke depression |
| 20000060 | Precerebral artery occlusion |
| 20000060 | Putamen haemorrhage |
| 20000060 | Quadriparesis |
| 20000060 | Quadriplegia |
| 20000060 | Red blood cells CSF positive |
| 20000060 | Reversible ischaemic neurological deficit |
| 20000060 | Ruptured cerebral aneurysm |
| 20000060 | Sneddon's syndrome |
| 20000060 | Spastic paralysis |

| SMQ Code | Preferred term |
|----------|-------------------------------------------------|
| 20000060 | Spastic paraplegia |
| 20000060 | Spinal artery embolism |
| 20000060 | Spinal artery thrombosis |
| 20000060 | Spinal cord haemorrhage |
| 20000060 | Spinal epidural haemorrhage |
| 20000060 | Spinal haematoma |
| 20000060 | Spinal vascular disorder |
| 20000060 | Spinal vessel congenital anomaly |
| 20000060 | Stroke in evolution |
| 20000060 | Subarachnoid haemorrhage |
| 20000060 | Subarachnoid haemorrhage neonatal |
| 20000060 | Subclavian steal syndrome |
| 20000060 | Subdural haematoma |
| 20000060 | Subdural haematoma evacuation |
| 20000060 | Subdural haemorrhage |
| 20000060 | Subdural haemorrhage neonatal |
| 20000060 | Superficial siderosis of central nervous system |
| 20000060 | Superior sagittal sinus thrombosis |
| 20000060 | Susac's syndrome |
| 20000060 | Thalamic infarction |
| 20000060 | Thalamus haemorrhage |
| 20000060 | Thrombotic cerebral infarction |
| 20000060 | Thrombotic stroke |
| 20000060 | Transient ischaemic attack |
| 20000060 | Transverse sinus thrombosis |
| 20000060 | Vascular encephalopathy |
| 20000060 | Vasculitis cerebral |
| 20000060 | Vertebral artery dissection |
| 20000060 | Vertebral artery occlusion |
| 20000060 | Vertebral artery stenosis |
| 20000060 | Vertebral artery thrombosis |
| 20000060 | Vertebrobasilar dolichoectasia |
| 20000060 | Vertebrobasilar insufficiency |
| 20000060 | Visual midline shift syndrome |
| 20000060 | Wallenberg syndrome |

# 10.3.3. Medical history of ischemic heart disease /Myocardial Infarction: defined by MSSO SMO 20000047

PBMQ 'Myocardial Infarction' is defined by selected PTs only (from MSSO SMQs below):

20000043: Ischaemic heart disease (MSSO SMQ)

20000047: Myocardial infarction (MSSO SMQ)

| Ischaemic heart disease (SMQ) | 20000043 | Acute coronary syndrome |
|---|---|---|
| Ischaemic heart disease (SMQ) | 20000043 | Acute myocardial infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Angina pectoris |
| Ischaemic heart disease (SMQ) | 20000043 | Angina unstable |
| Ischaemic heart disease (SMQ) | 20000043 | Arteriogram coronary abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Arteriosclerosis coronary artery |
| Ischaemic heart disease (SMQ) | 20000043 | Arteriospasm coronary |
| Ischaemic heart disease (SMQ) | 20000043 | Blood creatine phosphokinase MB abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Blood creatine phosphokinase MB increased |
| Ischaemic heart disease (SMQ) | 20000043 | Blood creatine phosphokinase abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Blood creatine phosphokinase increased |
| Ischaemic heart disease (SMQ) | 20000043 | Cardiac enzymes increased |
| Ischaemic heart disease (SMQ) | 20000043 | Cardiac stress test abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Computerised tomogram coronary artery abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary angioplasty |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary arterial stent insertion |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery bypass |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery disease |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery dissection |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery embolism |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery insufficiency |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery occlusion |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery reocclusion |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery restenosis |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery stenosis |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary artery thrombosis |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary bypass thrombosis |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary endarterectomy |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary no-reflow phenomenon |
| Ischaemic heart disease (SMQ) | 20000043 | Coronary ostial stenosis |

| Ischaemic heart disease (SMQ) | 20000043 | Coronary revascularisation |
|---|---|---|
| Ischaemic heart disease (SMQ) | 20000043 | Dissecting coronary artery aneurysm |
| Ischaemic heart disease (SMQ) | 20000043 | ECG electrically inactive area |
| Ischaemic heart disease (SMQ) | 20000043 | ECG signs of myocardial ischaemia |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram Q wave abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST segment abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST segment depression |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST segment elevation |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST-T segment abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST-T segment depression |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram ST-T segment elevation |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram T wave abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Electrocardiogram T wave inversion |
| Ischaemic heart disease (SMQ) | 20000043 | Exercise electrocardiogram abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Exercise test abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | External counterpulsation |
| Ischaemic heart disease (SMQ) | 20000043 | Haemorrhage coronary artery |
| Ischaemic heart disease (SMQ) | 20000043 | Infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Ischaemic cardiomyopathy |
| Ischaemic heart disease (SMQ) | 20000043 | Kounis syndrome |
| Ischaemic heart disease (SMQ) | 20000043 | Microvascular coronary artery disease |
| Ischaemic heart disease (SMQ) | 20000043 | Myocardial infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Myocardial ischaemia |
| Ischaemic heart disease (SMQ) | 20000043 | Myocardial reperfusion injury |
| Ischaemic heart disease (SMQ) | 20000043 | Myocardial stunning |
| Ischaemic heart disease (SMQ) | 20000043 | Papillary muscle infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Percutaneous coronary intervention |
| Ischaemic heart disease (SMQ) | 20000043 | Post procedural myocardial infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Postinfarction angina |
| Ischaemic heart disease (SMQ) | 20000043 | Prinzmetal angina |
| Ischaemic heart disease (SMQ) | 20000043 | Scan myocardial perfusion abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Silent myocardial infarction |
| Ischaemic heart disease (SMQ) | 20000043 | Stress cardiomyopathy |
| Ischaemic heart disease (SMQ) | 20000043 | Stress echocardiogram abnormal |
| Ischaemic heart disease (SMQ) | 20000043 | Subclavian coronary steal syndrome |

| | 1 | |
|---|---|---|
| Ischaemic heart disease (SMQ) | 20000043 | Subendocardial ischaemia |
| Ischaemic heart disease (SMQ) | 20000043 | Troponin I increased |
| Ischaemic heart disease (SMQ) | 20000043 | Troponin T increased |
| Ischaemic heart disease (SMQ) | 20000043 | Troponin increased |
| Ischaemic heart disease (SMQ) | 20000043 | Vascular graft occlusion |
| Medical history of myocardial infarction (aflibercept) | SMQ_1278 | Acute coronary syndrome |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Acute myocardial infarction |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Angina pectoris |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Angina unstable |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Arteriogram coronary abnormal |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Arteriosclerosis coronary artery |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Arteriospasm coronary |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Computerised tomogram coronary artery abnormal |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary angioplasty |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary arterial stent insertion |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery bypass |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery disease |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery dissection |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery embolism |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery insufficiency |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery occlusion |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery reocclusion |

| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery restenosis |
|---|---|---|
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery stenosis |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary artery thrombosis |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary bypass thrombosis |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary endarterectomy |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary no-reflow phenomenon |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary ostial stenosis |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Coronary revascularisation |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Dissecting coronary artery aneurysm |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | ECG electrically inactive area |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | ECG signs of myocardial ischaemia |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST segment abnormal |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST segment depression |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST segment elevation |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST-T segment abnormal |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST-T segment depression |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Electrocardiogram ST-T segment elevation |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | External counterpulsation |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Haemorrhage coronary artery |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Infarction |
| infarction (VEGF Trap-Eye) Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 SMQ_1278 SMQ_1278 SMQ_1278 SMQ_1278 SMQ_1278 | Electrocardiogram ST segment elevation Electrocardiogram ST-T segment abnormal Electrocardiogram ST-T segment depression Electrocardiogram ST-T segment elevation External counterpulsation Haemorrhage coronary artery |

| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Ischaemic cardiomyopathy |
|---|---|---|
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Ischaemic contracture of the left ventricle |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Kounis syndrome |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Myocardial infarction |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Myocardial ischaemia |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Myocardial reperfusion injury |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Myocardial stunning |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Papillary muscle infarction |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Percutaneous coronary intervention |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Post procedural myocardial infarction |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Postinfarction angina |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Prinzmetal angina |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Scan myocardial perfusion abnormal |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Silent myocardial infarction |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Stress cardiomyopathy |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Subclavian coronary steal syndrome |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Subendocardial ischaemia |
| Medical history of myocardial infarction (VEGF Trap-Eye) | SMQ_1278 | Vascular graft occlusion |

### 10.3.4. Renal Impairment

Renal impairment is defined by CRCL values.

Categories for renal impairment:

- CLCR >80ml/min (normal),
- CLCR >50-80ml/min (mild),
- CLCR >30-50 ml/min (moderate),
- CLCR <=30ml/min or 'requiring dialysis' (severe)

CLCR will be calculated using baseline values (creatinine, age, weight, sex) using the Cockcroft-Gault equation:

Males: CLCR = (140-age)\*body weight / (72\*creatinine)

Females: CLCR = (140-age)\*body weight\*0.85 / (72\*creatinine)

### 'Requiring dialysis' is defined by PT from

| MSSO SMQ | MSSO SMQ Code | Preferred term |
|---|---|---|
| renal impairment requiring dialysis | 10061102 | Dependence on enabling machine or device |
| renal impairment requiring dialysis | 10061105 | Dialysis |
| renal impairment requiring dialysis | 10018875 | Haemodialysis |
| enal impairment requiring dialysis 10034660 | | Peritoneal dialysis |

# 10.4. Calculation of confidence intervals using Mantel-Haenszel weighting scheme

The confidence intervals using the Mantel-Haenszel weighting scheme will be calculated according to the formulas given by Koch et al. (1990, p. 415 ff.)<sup>2</sup>, i.e. to compute confidence intervals for the difference in two binomial proportions obtained from a multicenter trial, we calculate a weighted difference and its associated variance using Mantel-Haenszel weighting scheme.

For a multicenter study with h 2x2 tables, the weighted difference is:

$$d = (\sum w_h(p_{he} - p_{hs}))/(\sum w_h)$$

where  $w_h = n_{he}n_{hs}/(n_{he}+n_{hs})$ 

and  $p_{he}$  = success rate for experimental treatment in stratum h

p<sub>hs</sub> = success rate for standard treatment in stratum h

 $n_{he}$  = number of patients under experimental treatment in stratum h

 $n_{hs}$  = number of patients under standard treatment in stratum h

The variance of the weighted difference is:

$$var(d) = (\sum w_h^2 (p_{hs}(1-p_{hs})/(n_{hs}-1) + p_{he}(1-p_{he})/(n_{he}-1)))/(\sum w_h)^2$$

A large sample approximation is used to compute the confidence interval:

$$CI = d \pm z_{\alpha/2} SQRT(var(d))$$

Where  $z_{\alpha}$  is the  $\alpha$  quantile of the standard normal distribution and SQRT is the square root function.

## 10.5. Criteria for Predefined Lab Abnormalities

| Parameter | PCSVs for phase 2/3 studies |
|---|---|
| Clinical chemistry | |
| ALT | By distribution analysis: > 3 ULN |
| AST | By distribution analysis: > 3 ULN |
| Alkaline Phosphatase | > 1.5 ULN |
| Total Bilirubin | > 1.5 ULN |
| Conjugated bilirubin | > 35% total bilirubin (when total bilirubin >1.5 ULN) |
| ALT and Total Bilirubin | ALT > 3 ULN and Total Bilirubin > 2 ULN |
| СРК | > 3 ULN |
| Creatinine | ≥ 150 µmol/L (Adults)<br>≥ 30% from baseline |
| Uric Acid | Hyperuricemia: >408 μmol/L<br>Hypouricemia: <120 μmol/L |
| Blood Urea Nitrogen | ≥ 17 mmol/L |
| Chloride | < 80 mmol/L<br>> 115 mmol/L |
| Sodium | ≤ 129 mmol/L<br>≥ 160 mmol/L |
| Potassium | < 3 mmol/L<br>≥ 5.5 mmol/L |
| Total Cholesterol | ≥ 7.74 mmol/L (3 g/L) |
| Triglycerides | ≥ 4.6 mmol/L (4 g/L) |
| Lipasemia | ≥ 3 ULN |
| Amylasemia | ≥ 3 ULN |
| Glucose - Hypoglycaemia - Hyperglycaemia | ≤ 3.9 mmol/L and < LLN<br>≥ 11.1 mmol/L (unfasted), ≥ 7 mmol/L (fasted) |

| Parameter | PCSVs for phase 2/3 studies |
|---|---|
| HbA1c | > 8 % |
| Albumin | ≤ 25 g/L |
| CRP | > 2 ULN or<br>> 10 mg/L (if ULN not provided) |
| Hematology | |
| WBC | < 3.0 GIGA/L (non-Black), < 2.0 GIGA/L (Black), ≥ 16.0 GIGA/L |
| Lymphocytes | > 4.0 GIGA/L |
| Neutrophils | < 1.5 GIGA/L (non-Black)<br>< 1.0 GIGA/L (Black) |
| Monocytes | > 0.7 GIGA/L |
| Basophils | > 0.1 GIGA/L |
| Eosinophils | > 0.5 GIGA/L or<br>> ULN if ULN ≥ 0.5 GIGA /L |
| Hemoglobin | Males : 115 g/L ( $\leq$ 7.14 mmol/L), $\geq$ 185 g/L (11.48 mmol/L)<br>Females : $\leq$ 95 g/L (5.9 mmol/L), $\geq$ 165 g/L (10.24 mmol/L)<br>Decrease from Baseline $\geq$ 20 g/L (1.24 mmol/L) |
| Hematocrit | Males : $\leq 0.37 \text{ v/v}, \geq 0.55 \text{ v/v}$<br>Females : $\leq 0.32 \text{ v/v}, \geq 0.5 \text{ v/v}$ |
| RBC | ≥ 6 TERA/L |
| Platelets | < 100 GIGA/L<br>≥ 700 GIGA/L |

### 10.6. Process to Derive Week 24 (Week 52) Data Cut-off

For Week 24 (Week 52) evaluations, a strategy for performing the data cut-off for the clinical database was developed, as described in the following:

### 10.6.1. Visit Dependent Data

All visit dependent data up to Week 24 (Week 52) [Visit 7 (Visit 11)] will be kept for the Week 24 (Week 52) analysis. All visit dependent data later than Week 24 (Week 52) [Visit 7 (Visit 11)] will not be included for the Week 24 (Week 52) analysis. Unscheduled visits with a date up to Week 24 (Week 52) [Visit 7 (Visit 11)] visit date will be kept for the Week 24 (Week 52) analysis data. If patients did not have Week 24 (Week 52) [Visit 7 (Visit 11)] visit date, unscheduled visit will be kept up to date of first injection + 168 days for the Week 24 (Week 52) analysis.

### 10.6.2. Visit Independent Data

Visit independent data (or event based data) include adverse events, concomitant/prior medication, and surgical/medical history.

# Patients that discontinued study prematurely before or at Week 24 (Week 52) [Visit 7 (Visit 11)]

These patients are defined as having their end of study CRF page filled, and have either:

- a dropout date earlier or equal to date of first injection + 168 (364) days or
- a dropout date earlier or equal to Week 24 (Week 52) visit date

For such patients, all event based records are kept in the clinical database for Week 24 (Week 52) analysis without any change.

#### Patients who stayed longer than Week 24 (Week 52) [Visit 7 (Visit 11)] in the study

These patients are the patients who did not discontinue study prematurely at/before Week 24 (Week 52) [Visit 7 (Visit 11)]. Therefore, these patients are either:

- still ongoing after Week 24 (Week 52) [Visit 7 (Visit 11)],
- discontinued the study prematurely, but were in the study for longer than Week 24 (Week 52) [Visit 7 (Visit 11)].

For such patients, the following will be applied:

All event records with a start date later than the date of the Week 24 (Week 52) [Visit 7 (Visit 11)] will be censored. This includes the case that the incomplete date is without any doubt later than the Week 24 (Week 52) visit date, e.g. Week 24 (Week 52) [Visit 7 (Visit 11)] is 10 April 2010 and the incomplete date is May 2010 or only 2011. If Week 24 (Week 52) visit date is missing, then date of first injection + 168 (364) days will be used instead below.

Records with a start date earlier or equal to the date of Week 24 (Week 52) (first injection + 168 (364) days if date of Week 24 (Week 52) is missing) will be kept (this includes incomplete dates when the incomplete date is earlier than the week 24 (week 52) date or in case of doubts,

e.g., Week 24 (visit 9) is 10 April 2010 and the incomplete date is March 2010, April 2010 or only 2010 or even a missing date, but several adaptions to the data will be made):

#### • Concomitant medication:

If a stop date is reported which is earlier than the date of Week 24 (Week 52) [Visit 7 (Visit 11)] (first injection + 168 (364) days if date of Week 24 (Week 52) is missing), the record will not be changed.

If a stop date is reported which is later than the date of Week 24 (Week 52) [Visit 7 (Visit 11)] (first injection + 168 (364) days if date of Week 24 (Week 52) is missing), the stop date will be set to missing and the variable CMONG will be set to 1 (yes).

#### • Adverse Events:

AEs with a start date on or after the date of the Week 24 (Week 52) [Visit 7 (Visit 11)] will be censored. Cut-off date will be first injection + 168 (364) days if date of Week 24 (Week 52) is missing.

If a stop date of adverse event is specified and earlier or equal to date of Week 24 (Week 52) [Visit 7 (Visit 11)] (first injection + 168 (364) days if date of Week 24 (Week 52) missing), then the record will not be changed.

If a stop date of adverse event is specified and later than the date of Week 24 (Week 52) [Visit 7 (Visit 11)] (first injection + 168 (364) days if date of Week 24 (Week 52) is missing), then the stop date will be deleted (set to missing) and the outcome of the adverse event (SAS variable AEOUT) will be set to missing.

If no stop date is specified and the outcome is either not yet reported (AEOUT is blank) or is reported (AEOUT" is 2-recovering/resolving, 4-not recovered/not resolved, 992-unknown), then the outcome will be set to missing (AEOUT is blank).

### • Surgeries:

All surgeries with a date of surgery later than Week 24 (Week 52) [Visit 7 (Visit 11)] date will be deleted

### 10.6.3. Study Medication Data

Study medication data (including real/sham injection) up to Week 16 (Week 48) [Visit 6 (Visit 10)] will be kept for the Week 24 (Week 52) analysis.

### 10.7. SAS Procedure for Multiple Imputation

<u>Step 1. Imputation:</u> Impute missing value using MCMC method and subsequently impute missing data by a regression model.

```
PROC MI DATA = <indata> SEED = 12345 OUT=mi01 NIMPUTE = 100; *SEED = 12345;

MCMC IMPUTE =MONOTONE;

VAR v1 v2 v3 v4 v5 ...;

RUN;

PROC MI DATA=mi01 SEED=54321 OUT= mi02 NIMPUTE=1;

CLASS <treatment> <factor>;

MONOTONE REG;

VAR <treatment> <factor> v1 v2 v3 v4 v5 ...;

BY _IMPUTATION_;

RUN;
```

<u>Step 2. Analysis:</u> After merge imputed data with the original data, define respond as ≥2 steps decrease from baseline in the DRSS score. Use PROC FREQ CMH to analyze data by \_imputation\_.

```
ODS OUTPUT CMH=cmh;

PROC FREQ DATA=<combined data>;

BY _IMPUTATION_;

TABLES <factor>*<treatment>*<respond>/CMH;

RUN;
```

### Step 3. Polling

Apply Wilson-Hilferty transformation to the CMH statistic and standardize the resulting normal variable. Then combine results and Compute one-sided p-value.

```
DATA cmh_wh;

SET cmh(WHERE=(AltHypothesis="General Association"));

cmh_value_wh=((VALUE/DF)**(1/3) - (1-2/(9*DF)))/SQRT(2/(9*DF));

cmh_sterr_wh = 1.0;

RUN;

ODS OUTPUT PARAMETERESTIMATES=mian_cmh_wh;

PROC MIANALYZE DATA=cmh_wh;

MODELEFFECTS cmh_value_wh;

STDERR cmh_sterr_wh;

RUN;

DATA pval (keep = PROBT_UPPER);

SET mian_cmh_wh;

IF tValue > 0 THEN Probt_upper = Probt/2;

ELSE Probt_upper = 1-Probt/2;

RUN;
```

### Signature Page for VV-RIM-00052364 v1.0



Signature Page for VV-RIM-00052364 v1.0 Approved